CLINICAL TRIAL: NCT04853706
Title: Validation of the 3D-CAM Turkish Version in Surgical ICU Patients
Brief Title: Validation of the 3D-CAM Turkish Version
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SINEM SARI, Assoc Prof, Aydin Adnan Menderes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021/28
Record Dates: First submitted 2021-04-13; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Delirium; Validity
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Delirium (Other)
  Interventions: Diagnostic Test: 3d cam; Diagnostic Test: DSM 5

INTERVENTIONS:
Diagnostic Test: 3d cam — The 3D-CAM is a short interview that uses verbal responses and allows completion of the Confusion Assessment Method (CAM) diagnostic algorithm
Diagnostic Test: DSM 5 — The DSM-5 is the gold standard for diagnosing delirium. But proper use requires professional psychiatric background and training.

SUMMARY:
3D CAM into Turkish validity and reliability on postoperative delirium will be test as a prospective diagnostic study. After approval by Dr. Edward R. Marcantonio, (15) will translation and back-translation. The original 3D-CAM will translate into Turkish by two medical doctor .The two translational versions will be discussed and merged into a final version. Back translation will performed in regardless of any information from its original version by another two medical doctor. Both the translated and back translated versions will sent to Dr. Marcantonio for approval. Eligibility and the documentation of consent will be confirmed at the preoperative visit. During this visit, patients will provide demographic and historical medical information, including information regarding medication usage. The Mini-Mental State Exam (MMSE) will be performed.

Delirium assessment

Delirium assessment with the 3D-CAM Before the study period, all researchers will participate online training program on 3D CAM. Delirium will be evaluated using the 3D CAM every each morning and evening (18:00-20:00) for postoperative 3 days.

Delirium assessment with the DSM-5 The psychiatrist investigator who was blinded to the 3D-CAM assessment results, will evaluate the patients according to the criteria of DSM-5 within 3 min after the 3D-CAM assessment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* ASA Physical Status 1-3
* Admitted to the ICU after surgery with a predicted length of stay for more than 48 h
* MMSE ≥ 20 (to exclude dementia)

Exclusion Criteria:

* Refused to participate
* Patients with severe visual or auditory disorder/handicaps or endotracheal intubation which might impede communication
* Presence of a major psychiatric condition such as bipolar disorder, major depression, schizophrenia, Alzheimer or dementia, Parkinsonism
* Deep sedation or coma
* ASA physical status IV or V

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2021-04-18 (Estimated); Primary Completion 2021-10-18 (Estimated); Study Completion 2021-12-18 (Estimated)

PRIMARY OUTCOMES:
Assessment of delirium | 3 days
  Delirium will be evaluated using the 3D CAM every each morning and evening (18:00-20:00) for postoperative 3 days. The psychiatrist investigator who will be blinded to the 3D-CAM assessment results, will evaluate the patients according to the criteria of DSM-5 within 3 min after the 3D-CAM assessment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mu DL, Ding PP, Zhou SZ, Liu MJ, Sun XY, Li XY, Wang DX. Cross-cultural adaptation and validation of the 3D-CAM Chinese version in surgical ICU patients. BMC Psychiatry. 2020 Mar 24;20(1):133. doi: 10.1186/s12888-020-02544-w. PMID 32204700